CLINICAL TRIAL: NCT02489448
Title: Single Arm Neoadjuvant Phase I/II Study of MEDI4736 (Anti-PD-L1 Antibody) Concomitant With Weekly Nab-paclitaxel and Dose-dense Doxorubicin/Cyclophosphamide (ddAC) Chemotherapy for Clinical Stage I-III Triple Negative Breast Cancer
Brief Title: Neoadjuvant MEDI4736 Concomitant With Weekly Nab-paclitaxel and Dose-dense AC for Stage I-III Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1409014537
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEDI4736 (Experimental): The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736 — The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
  Other Names: tremelimumab, anti-PD-L1 antibody

SUMMARY:
The purpose of the study is to address the following hypotheses: (i) Anti-PD-L1 therapy with MEDI4736 administered concomitantly with weekly nab-paclitaxel followed by MEDI4736 concomitant with ddAC neoadjuvant chemotherapy will induce higher pathologic complete response (pCR) rate (>55%) in triple negative breast cancer than historical pCR rates (30-40%) observed with chemotherapy alone. (ii) MEDI4736 can be safely co-administered at full dose with sequential with nab-paclitaxel (100mg/m2) and ddAC (60 mg/m2 and 600 mg/m2 respectively).

DETAILED DESCRIPTION:
The primary objective of the Phase I portion of the trial is to assess the safety of MEDI4736 combined with chemotherapy and determine if full dose of MEDI4736 can be administered concomitantly with full dose weekly nab-paclitaxel followed by dose-dense AC chemotherapies, respectively.

The primary objective of the Phase II portion of the study is to estimate the pCR rate with MEDI4736 in combination with weekly nab-paclitaxel x 12 treatments followed by MEDI4736 in combination with ddAC x 4 treatments for estrogen receptor (ER), progesterone receptor (PR) and HER2 negative (triple negative, TNBC), clinical stage I-III breast cancer. Pathologic complete response is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e. ypT0/Tis ypN0).

Secondary objectives include: to assess the safety and toxicity of adding anti-PD-L1 antibody, MEDI4736 to standard of care neoadjuvant chemotherapy in the Phase II portion of the trial. The study will also monitor for events of special clinical interest with a suspected auto-immunologic etiology including grade ≥3 colitis, hyperthyroidism, hypophysitis, hypothyroidism, pneumonitis, rash and anti-drug-antibody (ADA) immune complex disease (manifested by symptoms of arthralgias, abdominal pain, back pain, and vasculitis).

Exploratory objectives include: to assess correlation between response to therapy and immune parameters of the tumor at baseline and post-treatment in patients who have residual cancer after therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically confirmed stage I-III, ER, PR and HER2 negative invasive breast cancer as defined by the ASCO CAP guidelines for whom systemic chemotherapy would be indicated based on physician judgment following standard NCCN practice guidelines.
2. Willing and able to provide written informed consent for voluntary participation in the trial.
3. Willing to undergo a baseline tumor core needle biopsy and blood draws for correlative science studies.
4. Eighteen years of age or older on the day of signing informed consent.
5. Female subjects must either be of non-reproductive potential or must have a negative urine or serum pregnancy test upon study entry.
6. Patients should have adequate organ function to tolerate chemotherapy, as defined by:

   * peripheral granulocyte count of > 1,500/mm3
   * platelet count > 100,000/mm3
   * hemoglobin >9 g/dL
   * total bilirubin < 1.5 x upper limit of normal (ULN)
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) each < 1.5 x ULN
   * serum creatinine < 1.5 x ULN or serum creatinine clearance < 50mL/min
   * INR/PT/PTT each < 1.5 x ULN
   * TSH within normal limits

Exclusion Criteria:

1. Patients who underwent partial excisional biopsy or lumpectomy, segmental mastectomy or modified radical mastectomy or sentinel node.
2. Patients for whom anthracycline, paclitaxel or antibody therapies are contraindicated.
3. Patients with active autoimmune disease or documented autoimmune disease within 2 years. Patients with hypothyroidism that is clinically stable and have normal TSH levels with hormone replacement, or patients with vitiligo or psoriasis not requiring treatment remain eligible for the study.
4. Active or prior documented inflammatory bowel disease (Crohn's disease, ulcerative colitis).
5. Patients with known active hepatitis B or C or HIV infection or with history of tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11; Primary Completion 2021-06-15 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, D. Phil., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 patients took part in the Phase 1 portion of the study. 61 patients took part in the Phase 2 portion of this study, for which results are presented. 2 removed consent once placed on study.
Groups:
- MEDI4736: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
  MEDI4736: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
Period: Overall Study
Arm/Group | MEDI4736
Started | 68
Phase 1 Started | 7
3 mg Dose | 4
10 mg Dose | 3
Phase 1 Completed | 7
Phase 2 Started | 61
Phase 2 Completed | 56 (56 phase 2 patients had surgery to be assessed for the primary outcome.)
Completed | 63 (The total comes from: 7 Phase 1 patients and 56 Phase 2 patients with surgery to be assessed for the primary outcome. 5 Phase 2 patients did not complete the study.)
Not Completed | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Patients enrolled in Phase 2, 2 of 61 removed consent and withdrew, they are not presented here in the results (baseline characteristics and primary outcome) but were counted in the adverse events.
Groups:
- Phase 1: 3mg MEDI4736; Phase 1: 10mg MEDI4736; Phase 2: 10mg MEDI4736: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
  MEDI4736: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 3mg MEDI4736 | Phase 1: 10mg MEDI4736 | Phase 2: 10mg MEDI4736 | Total
Number analyzed (Participants) | 4 | 3 | 59 | 66
Age, Continuous [Median (Full Range); unit: years] | 56 [43 to 60] | 50 [40 to 54] | 51 [27 to 79] | 51.5 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 59 | 66
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White (non-Hispanic) | 4 | 2 | 35 | 41
  Race/Ethnicity: Hispanic/Latino | 0 | 1 | 5 | 6
  Race/Ethnicity: Black | 0 | 0 | 11 | 11
  Race/Ethnicity: Asian/American Indian | 0 | 0 | 4 | 4
  Race/Ethnicity: Unknown | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 59 | 66

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: Pathologic response will be assessed in the surgically resected cancer and lymph nodes after completion of all chemotherapy by the local pathologist as part of routine care. Pathologic complete response is defined as no invasive cancer in the resected breast tissue and lymph nodes (ypT0/Tis, ypN0).
  The outcome was changed from 19 weeks at the time of results entry as the treatment period was actually 20 weeks and the outcome was assessed 4-6 weeks after treatment when surgery took place.
Time Frame: Up to 26 weeks
Population: 56 of 59 patients had surgery performed
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 56
Participants | 25

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: Adverse events are reported for Phase 1 doses combined and Phase 2. At the time of data collection in Phase 1, adverse events were collected at the patient level, not at the dosing level.
Groups:
- Phase 1: MEDI4736 3mg & 10mg; Phase 2: MEDI4736 10mg: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
  MEDI4736: The investigational product is MEDI4736 which will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.
  Routine, standard of care chemotherapy will be given together with the investigational product and will include weekly nab-paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments.
Arm/Group | Phase 1: MEDI4736 3mg & 10mg | Phase 2: MEDI4736 10mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 3/61
Serious Adverse Events (participants affected / at risk) | 3/7 | 23/61
Other Adverse Events (participants affected / at risk) | 7/7 | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: MEDI4736 3mg & 10mg (N=7) | Phase 2: MEDI4736 10mg (N=61)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 3 (3)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify - Community Acquired Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Investigations - Other, specify - Diverticulitis (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify - Altered mental status. (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify - Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify - UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify - Skin and subcutaneous tissue disorders- Ot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (3)
Vascular disorders - Other, specify - Labile BP (SBP 50s - 190s). (Vascular disorders) | 0 (0) | 1 (2)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: MEDI4736 3mg & 10mg (N=7) | Phase 2: MEDI4736 10mg (N=61)
Nausea (Gastrointestinal disorders) | 5 (9) | 43 (68)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 28 (44)
Constipation (Gastrointestinal disorders) | 3 (4) | 26 (31)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 22 (25)
Vomiting (Gastrointestinal disorders) | 2 (3) | 15 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 9 (10)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 8 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 47 (67)
Headache (Nervous system disorders) | 2 (2) | 28 (35)
Dysgeusia (Nervous system disorders) | 5 (6) | 22 (23)
Dizziness (Nervous system disorders) | 2 (2) | 18 (24)
Paresthesia (Nervous system disorders) | 0 (0) | 13 (15)
Presyncope (Nervous system disorders) | 0 (0) | 5 (7)
Sinus pain (Nervous system disorders) | 0 (0) | 4 (4)
Fatigue (General disorders) | 5 (8) | 46 (82)
Pain (General disorders) | 3 (4) | 7 (8)
Non-cardiac chest pain (General disorders) | 1 (1) | 8 (8)
Fever (General disorders) | 0 (0) | 6 (6)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 6 (7)
Edema limbs (General disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 42 (52)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4) | 23 (32)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 21 (35)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 14 (16)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 11 (12)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 15 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 13 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5)
Musculoskeletal and connective tissue disorder - Other, (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 18 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 17 (24)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (9)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Watering eyes (Eye disorders) | 4 (4) | 12 (12)
Blurred vision (Eye disorders) | 2 (2) | 10 (10)
Dry eye (Eye disorders) | 1 (1) | 5 (5)
Eye disorders - Other (Eye disorders) | 1 (2) | 5 (6)
Lymphocyte count decreased (Investigations) | 0 (0) | 12 (24)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 11 (19)
Neutrophil count decreased (Investigations) | 0 (0) | 11 (24)
Alanine aminotransferase increased (Investigations) | 0 (0) | 10 (17)
White blood cell decreased (Investigations) | 0 (0) | 9 (24)
Weight loss (Investigations) | 0 (0) | 8 (9)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (6)
Platelet count decreased (Investigations) | 0 (0) | 5 (6)
Investigations - Other (Investigations) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 18 (22)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 9 (12)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 7 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 6 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Upper respiratory infection (Infections and infestations) | 2 (3) | 7 (9)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 7 (13)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 26 (73)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Hot flashes (Vascular disorders) | 4 (4) | 11 (11)
Hypertension (Vascular disorders) | 0 (0) | 12 (33)
Flushing (Vascular disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 20 (23)
Depression (Psychiatric disorders) | 0 (0) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (5)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 12 (14)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 9 (10)
Hematuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 4 (5)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 6 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (6)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 5 (6)
Floaters (Eye disorders) | 2 (3) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02489448/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02489448/SAP_001.pdf